CLINICAL TRIAL: NCT04575662
Title: Linac Based STereotactic Arrhythmia Radioablation (STAR) of Atrial Fibrillation
Brief Title: Radiotherapy and Atrial Fibrillation
Acronym: STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Massimo Grimaldi, Head of Arrhythmology and Electrophysiology Unit, Miulli General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGH_002
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Rhythm Control Strategy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: STAR treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAR Treatment (Experimental): Patients performing STAR treatment
  Interventions: Radiation: STAR Treatment

INTERVENTIONS:
Radiation: STAR Treatment — Radiation therapy that delivers non-invasive, image-guided, precise high-dose of radiation to targets reducing dose exposure to adjacent normal tissue and minimizing the treatment toxicity.

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia. Current European guidelines recommend catheter ablation of AF in symptomatic patients refractory to antiarrhythmic therapy. Pulmonary vein isolation (PVI) remains the cornerstone of any ablation procedure irrespective of patient characteristics. Recently, stereotactic arrhythmia radioablation (STAR) with precise high-dose of radiation was used to treat ventricular arrhythmias in patients with a high risk of complications during transcatheter ablation.

DETAILED DESCRIPTION:
Exploratory study to investigate the feasibility of STAR for the treatment of paroxysmal AF in elderly patients in which a rhythm control strategy is indicated. Patients will be followed-up for 12 months after STAR treatment for a safety assessment and AF recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 70 years
2. Symptomatic Paroxysmal AF
3. Antiarrhythmic drugs intolerance or non-response to antiarrhythmic drugs
4. Understands the nature of the study, treatment procedure and provides written informed consent
5. Willing to comply with specified pre-, post- and follow-up testing, evaluations and requirements
6. Expected to remain available for at least 24 months after enrollment

Exclusion Criteria:

1. Permanent AF
2. Need or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
3. Unstable angina
4. Presence of any disease that is likely to shorten life expectancy to < 1 year
5. Any cardiac surgery within three months prior to enrolment
6. Awaiting cardiac transplantation or other cardiac surgery within the next year
7. Myocardial infarction (MI) within 60 days prior to enrolment
8. Contraindications to oral anticoagulation
9. Active systemic infection or sepsis
10. Left atrial thrombus (e.g., transesophageal echocardiogram (TEE), CT and ICE)
11. History of a documented thromboembolic event such as stroke or transient ischemic neurological attack (TIA) in the three months prior to enrollment.
12. Currently enrolled in another trial that has not completed the required follow-up period and would conflict with this study.
13. Any other clinical condition that might jeopardize patient safety during participation in this trial or prevent the subject from adhering to the trialprotocol

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events related to STAR treatment | Baseline through 12-months
  To estimate the cumulative proportion of patients' Adverse Events related to STAR treatment

SECONDARY OUTCOMES:
Incidence of AF recurrence | Baseline through 12-months
  To estimate the proportion of patients with AF
Long-term clinical outcomes | Baseline through 10-years
  To estimate the cumulative proportion of all-cause death, cardiovascular death, stroke, heart failure hospitalization, AF recurrence, cancer occurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Miulli General Hospital, Acquaviva delle Fonti, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Monaco A, Gregucci F, Bonaparte I, Romanazzi I, Troisi F, Surgo A, Vitulano N, Quadrini F, Valenti N, Carbonara R, Di Guglielmo FC, Ludovico E, Calbi R, Guida P, Ciliberti MP, Fiorentino A, Grimaldi M. Linear accelerator-based stereotactic arrhythmia radioablation for paroxysmal atrial fibrillation in elderly: a prospective phase II trial. Europace. 2023 Dec 6;25(12):euad344. doi: 10.1093/europace/euad344. PMID 37988294
- [Derived] Di Monaco A, Gregucci F, Bonaparte I, Troisi F, Surgo A, Di Molfetta D, Vitulano N, Quadrini F, Carbonara R, Ludovico E, Ciliberti MP, Fiorentino A, Grimaldi M. First Pulmonary Vein Isolation Using LINAC-Based STAR. Circ Arrhythm Electrophysiol. 2022 Jun;15(6):e010880. doi: 10.1161/CIRCEP.122.010880. Epub 2022 Jun 1. No abstract available. PMID 35649117
- [Derived] Di Monaco A, Gregucci F, Bonaparte I, Troisi F, Surgo A, Di Molfetta D, Vitulano N, Quadrini F, Carbonara R, Martinelli G, Guida P, Ciliberti MP, Fiorentino A, Grimaldi M. Paroxysmal Atrial Fibrillation in Elderly: Worldwide Preliminary Data of LINAC-Based Stereotactic Arrhythmia Radioablation Prospective Phase II Trial. Front Cardiovasc Med. 2022 Mar 2;9:832446. doi: 10.3389/fcvm.2022.832446. eCollection 2022. PMID 35310997